CLINICAL TRIAL: NCT01169493
Title: Pacing Affects Cardiovascular Endpoints in Patients With Right Bundle-Branch Block (The PACE-RBBB Trial)
Acronym: PACE-RBBB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00025144; 10CRP3630033 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Heart Failure; Right Bundle-Branch Block
Keywords: Heart Failure; Right Bundle-Branch Block; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- VVI-40 to RV DDD-40 to Bi-V DDD-40 (Experimental): Period 1: Participants assigned to VVI-40 Participants will then Crossover to Period 2. Period 2: Participants assigned to RV DDD-40 Participants will then Crossover to Period 3. Period 3: Participants assigned to Bi-V DDD-40
  Interventions: Device: VVI-40; Device: RV DDD-40; Device: BiV DDD-40
- VVI-40 to Bi-V DDD-40 to RV DDD-40 (Experimental): Period 1: Participants assigned to VVI-40 Participants will then Crossover to Period 2. Period 2: Participants assigned to Bi-V DDD-40 Participants will then Crossover to Period 3. Period 3: Participants assigned to RV DDD-40
  Interventions: Device: VVI-40; Device: RV DDD-40; Device: BiV DDD-40
- Bi-V DDD-40 to VVI-40 to RV DDD-40 (Experimental): Period 1: Participants assigned to Bi-V DDD-40 Participants will then Crossover to Period 2. Period 2: Participants assigned to VVI-40 Participants will then Crossover to Period 3. Period 3: Participants assigned to RV DDD-40
  Interventions: Device: VVI-40; Device: RV DDD-40; Device: BiV DDD-40
- Bi-V DDD-40 to RV DDD-40 to VVI-40 (Experimental): Period 1: Participants assigned to Bi-V DDD-40 Participants will then Crossover to Period 2. Period 2: Participants assigned to RV DDD-40 Participants will then Crossover to Period 3. Period 3: Participants assigned to VVI-40
  Interventions: Device: VVI-40; Device: RV DDD-40; Device: BiV DDD-40
- RV DDD-40 to VVI-40 to Bi-V DDD-40 (Experimental): Period 1: Participants assigned to RV DDD-40 Participants will then Crossover to Period 2. Period 2: Participants assigned to VVI-40 Participants will then Crossover to Period 3. Period 3: Participants assigned to Bi-V DDD-40
  Interventions: Device: VVI-40; Device: RV DDD-40; Device: BiV DDD-40
- RV DDD-40 to Bi-V DDD-40 to VVI-40 (Experimental): Period 1: Participants assigned to RV DDD-40 Participants will then Crossover to Period 2. Period 2: Participants assigned to Bi-V DDD-40 Participants will then Crossover to Period 3. Period 3: Participants assigned to VVI-40
  Interventions: Device: VVI-40; Device: RV DDD-40; Device: BiV DDD-40

INTERVENTIONS:
Device: VVI-40 — Pacing mode set to VVI-40, RV only pacing
Device: RV DDD-40 — ICD programmed to DDD-40, RV only pacing with aan AV interval producing QRS fusion on surface EKG.
Device: BiV DDD-40 — ICD programmed to BiV pacing at a lower rate of 40

SUMMARY:
Heart failure (HF) affects 5 million Americans and is responsible for more health-care expenditure than any other medical diagnosis. Approximately half of all HF patients have electrocardiographic prolongation of the QRS interval and ventricular dyssynchrony, a perturbation of the normal pattern of ventricular contraction that reduces the efficiency of ventricular work. Ventricular dyssynchrony is directly responsible for worsening HF symptomatology in this subset of patients. Resynchronization of ventricular contraction is usually achieved through simultaneous pacing of the left and right ventricles using a biventricular (BiV) pacemaker or implantable cardioverter-defibrillator. Clinical trial evidence supporting the use of BiV pacing in patients with prolonged QRS duration was obtained almost exclusively in patients with a left bundle-branch block (LBBB) electrocardiographic pattern. Recent evidence suggests that resynchronization of ventricular contraction in patients with LBBB can be obtained by univentricular left ventricular pacing with equal or superior clinical benefits compared to BiV pacing. Animal studies suggest that ventricular resynchronization can be obtained in subjects with right bundle-branch block (RBBB) through univentricular right ventricular pacing. No clinical trial evidence exists to support the use of BiV pacing in patients with RBBB. Thousands of patients with symptomatic HF and RBBB currently have univentricular ICDs in place for the prevention of sudden cardiac death. Most of these devices are currently programmed to avoid RV pacing. We aim to determine if ventricular resynchronization delivered through univentricular RV pacing improves symptoms in patients with RBBB and moderate to severe HF who have previously undergone BiV ICD implantation for symptomatic heart failure. We further aim to determine if ventricular resynchronization improves myocardial performance and ventricular geometry as detected by echocardiographic measures and quality of life for patients with HF and RBBB. We hypothesize that RV univentricular pacing delivered with an atrio-ventricular interval that maximizes ventricular synchrony is equivalent to BiV pacing for improvement in cardiac performance, HF symptoms, and positive ventricular remodeling in patients with HF and RBBB.

ELIGIBILITY:
Inclusion Criteria:

* Cardiomyopathy of either idiopathic or ischemic etiology
* NYHA class III, or IV symptoms
* Sinus rhythm
* QRS complex duration > 130 msec in ≥ 2 surface ECG leads with RBBB
* PR interval > 150 msec and < 240 msec
* Prior implantation of dual chamber BiV ICD with apical RV lead location

Exclusion Criteria:

* Myocardial infarction, major surgical procedure, or acute cardiac failure crisis requiring inotropes within 6 months of entry into the study
* Atrial fibrillation or flutter lasting >12 hours within the last 6 months
* Sick sinus syndrome, complete heart block, or other arrhythmias requiring pacemaker support
* Pregnancy
* Any other known condition other than heart failure that could limit exercise time or survival to < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Atwater, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- VVI-40 to RV DDD-40 to Bi-V DDD-40: Period 1: Participants assigned to VVI-40 Participants will then Crossover to Period 2.
  Period 2: Participants assigned to RV DDD-40 Participants will then Crossover to Period 3.
  Period 3: Participants assigned to Bi-V DDD-40
  VVI-40: Pacing mode set to VVI-40, RV only pacing
  RV DDD-40: ICD programmed to DDD-40, RV only pacing with aan AV interval producing QRS fusion on surface EKG.
  BiV DDD-40: ICD programmed to BiV pacing at a lower rate of 40
- VVI-40 to Bi-V DDD-40 to RV DDD-40: Period 1: Participants assigned to VVI-40 Participants will then Crossover to Period 2.
  Period 2: Participants assigned to Bi-V DDD-40 Participants will then Crossover to Period 3.
  Period 3: Participants assigned to RV DDD-40
  VVI-40: Pacing mode set to VVI-40, RV only pacing
  RV DDD-40: ICD programmed to DDD-40, RV only pacing with aan AV interval producing QRS fusion on surface EKG.
  BiV DDD-40: ICD programmed to BiV pacing at a lower rate of 40
- Bi-V DDD-40 to VVI-40 to RV DDD-40: Period 1: Participants assigned to Bi-V DDD-40 Participants will then Crossover to Period 2.
  Period 2: Participants assigned to VVI-40 Participants will then Crossover to Period 3.
  Period 3: Participants assigned to RV DDD-40
  VVI-40: Pacing mode set to VVI-40, RV only pacing
  RV DDD-40: ICD programmed to DDD-40, RV only pacing with aan AV interval producing QRS fusion on surface EKG.
  BiV DDD-40: ICD programmed to BiV pacing at a lower rate of 40
Period: Period 1 (6 Months)
Arm/Group | VVI-40 to RV DDD-40 to Bi-V DDD-40 | VVI-40 to Bi-V DDD-40 to RV DDD-40 | Bi-V DDD-40 to VVI-40 to RV DDD-40 | Bi-V DDD-40 to RV DDD-40 to VVI-40 | RV DDD-40 to VVI-40 to Bi-V DDD-40 | RV DDD-40 to Bi-V DDD-40 to VVI-40
Started | 2 | 4 | 5 | 0 | 0 | 5
Completed | 2 | 3 | 3 | 0 | 0 | 2
Not Completed | 0 | 1 | 2 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 0 | 3
Period: Period 2 (6 Months)
Arm/Group | VVI-40 to RV DDD-40 to Bi-V DDD-40 | VVI-40 to Bi-V DDD-40 to RV DDD-40 | Bi-V DDD-40 to VVI-40 to RV DDD-40 | Bi-V DDD-40 to RV DDD-40 to VVI-40 | RV DDD-40 to VVI-40 to Bi-V DDD-40 | RV DDD-40 to Bi-V DDD-40 to VVI-40
Started | 2 | 3 | 3 | 0 | 0 | 2
Completed | 2 | 3 | 3 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (6 Months)
Arm/Group | VVI-40 to RV DDD-40 to Bi-V DDD-40 | VVI-40 to Bi-V DDD-40 to RV DDD-40 | Bi-V DDD-40 to VVI-40 to RV DDD-40 | Bi-V DDD-40 to RV DDD-40 to VVI-40 | RV DDD-40 to VVI-40 to Bi-V DDD-40 | RV DDD-40 to Bi-V DDD-40 to VVI-40
Started | 2 | 3 | 3 | 0 | 0 | 2
Completed | 2 | 1 | 2 | 0 | 0 | 2
Not Completed | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VVI-40 to RV DDD-40 to Bi-V DDD-40 | VVI-40 to Bi-V DDD-40 to RV DDD-40 | Bi-V DDD-40 to VVI-40 to RV DDD-40 | Bi-V DDD-40 to RV DDD-40 to VVI-40 | RV DDD-40 to VVI-40 to Bi-V DDD-40 | RV DDD-40 to Bi-V DDD-40 to VVI-40 | Total
Number analyzed (Participants) | 2 | 4 | 5 | 0 | 0 | 5 | 16
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 |  |  | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 |  |  | 2 | 3
  >=65 years | 2 | 3 | 5 |  |  | 3 | 13
Gender [Number; unit: participants]
  Female | 0 | 0 | 0 |  |  | 0 | 0
  Male | 2 | 4 | 5 |  |  | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of the Trial Will be a Comparison of the Proportion of Patients in Each of the Three Treatment Groups Who Demonstrate Positive LV Remodeling, Defined as a Decrease in LV End Systolic Diameter of >5mm.
Time Frame: 6 months
Population: All participants who completed the six month period for VVI-40, RV DDD-40, Bi-V DDD-40 regardless of which arm they are randomized to. Participants may be counted as completing more than one period.
Measure: Number; unit: percentage of participants
Groups:
- VVI-40: The VVI-40 arm will be programmed to VVI (inhibited) mode at a lower rate of 40.
- RV DDD-40: RV DDD-40 will have an AV interval set to produce QRS fusion with the native conduction down the native left bundle
- Bi-V DDD-40: Permits direct comparison of RV univentricular pacing and current standard of care (BiV) pacing.
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 10 | 7 | 10
percentage of participants | 0 | 29 | 20

2. Secondary Outcome: Secondary Echocardiographic Endpoints
Description: Comparisons of the derived velocity-time integral calculated on the aortic continuous wave Doppler-spectrogram, RV end-diastolic size, RV EF, mitral and tricuspid regurgitation severity, and estimated RV systolic pressure.
Time Frame: 6 months
Population: Data not collected.
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Arrhythmic Events
Description: To determine if pacing mode impacts the frequency of ventricular arrhythmias, the incidence of ventricular tachyarrhythmia episodes on device interrogation will be compared between treatment group assignments. An episode will be considered ventricular arrhythmia if it lasts longer than 30 seconds or requires anti-tachycardia pacing or high voltage device therapy for termination.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 10 | 7 | 10
participants | 0 | 0 | 0

4. Secondary Outcome: Minnesota Quality of Life Questionnaire
Description: This is a standardized method for assessing quality of life in patients with heart failure. It asks 21 questions and measures the impact HF has on a subject's life. Each question is rated 0-5. The total score for the 21 items can range from 0 to 105. Higher scores indicate more burden of disease on quality of life.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 10 | 7 | 10
units on a scale | 39.3 (21.3) | 43.9 (20.3) | 55.78 (27.7)

5. Secondary Outcome: 6-minute Walk Distance
Description: 6-minute walk distance was the distance that a participant could walk in 6 minutes.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 10 | 7 | 10
meters | 292.4 (70.5) | 235.8 (122.8) | 244.44 (122)

6. Secondary Outcome: NYHA Function Class
Description: The New York Heart Association (NYHA) Functional Classification places patients in one of four categories based on how much they are limited during physical activity. Class I means there is no limitation of physical activity and Class IV means a person is unable to carry on any physical activity without discomfort/symptoms of heart failure at rest.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 10 | 7 | 10
units on a scale | 3.3 (0.7) | 3 (0.6) | 3.2 (0.9)

7. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 6 months
Population: Data not collected.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 10 | 7 | 10
percent | 24.8 (7.4) | 20 (9.7) | 22.9 (7.7)

8. Secondary Outcome: Left Ventricular End-diastolic Size
Time Frame: 6 months
Population: Data not collected.
Measure: Mean (Standard Error); unit: cubic cm
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Number analyzed (Participants) | 10 | 7 | 10
cubic cm | 203 (39.9) | 236.6 (27.1) | 236.5 (54.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 18 months
Groups:
- RV DDD-40: RV DDD-40: ICD programmed to DDD-40, RV only pacing with an AV interval producing QRS fusion on surface EKG.
- Bi-V DDD-40: Bi-V DDD-40: ICD programmed to Bi-V pacing at a lower rate of 40
Arm/Group | VVI-40 | RV DDD-40 | Bi-V DDD-40
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 3/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VVI-40 (N=11) | RV DDD-40 (N=13) | Bi-V DDD-40 (N=12)
Heart Failure Exacerbation, Heart Transplant (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Death (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We were unable to enroll adequately, and the study was underpowered to assess either the safety or efficacy of RV only, or BIV pacing in patients with right bundle branch block.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No